CLINICAL TRIAL: NCT00407056
Title: Phase 3 Open-Labeled Study of 0.05% Difluprednate Ophthalmic Emulsion in the Treatment of Severe Anterior Uveitis (Including Panuveitis).
Brief Title: Study of Difluprednate Ophthalmic Emulsion in the Treatment of Severe Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJE2079/3-02-PC
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Uveitis; Panuveitis
MeSH Terms: conditions — Uveitis; Panuveitis

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion

SUMMARY:
The purpose of this phase 3 open-labeled study is to determine if difluprednate ophthalmic emulsion is effective in the treatment of severe uveitis.

DETAILED DESCRIPTION:
The objective of this phase 3 study is to assess the efficacy and safety of 0.05% difluprednate ophthalmic emulsion in patients with severe endogenous anterior uveitis with an open-labeled, no-controlled and no-randomized design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of endogenous anterior uveitis or panuveitis
* Patients with ≥ 50 anterior chamber cells as observed by slit lamp microscopy (criterion for evaluation of signs 4)
* Patients requiring more frequent instillation of 0.1% betamethasone sodium phosphate ophthalmic solution than the regular frequency specified in its dosage and administration (3 - 4 times/day)
* Patients aged ≥ 12 years (on the day of obtaining informed consent) who were able to actuate symptoms
* Patients giving written informed consent prior to initiation of the study

Exclusion Criteria:

* Patients who did not meet all of the above inclusion criteria
* Patients initiating treatment with systemic administration of any corticosteroid, non-steroidal anti-inflammatory drug, antiphlogistic enzyme or immunosuppressive drug within 2 weeks before instillation of the investigational drug
* Patients receiving topical injection of any corticosteroid in eyes before instillation of the investigational product(solution formulation: within 1 week before instillation of the investigational product, depot formulation: within 2 weeks before instillation of the investigational product)
* Patients receiving instillation of any corticosteroid, non-steroidal anti-inflammatory ophthalmic solution or antiphologistic enzyme within 12 hours before instillation of the investigational drug
* Patients with glaucoma or ocular hypertension
* Patients with corneal erosion or corneal ulcer
* Patients with any viral, bacterial or fungal keratoconjunctival disease or suspected with eye infection
* Patients with allergy to similar drugs of difluprednate
* Patients requiring use of contact lens during the study period
* Women who were or might be pregnant, or lactating women
* Patients participating in another clinical study within 3 months before initiation of the present study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2002-08; Study Completion 2003-06

PRIMARY OUTCOMES:
The anterior chamber cell score was compared between baseline and Day 14.

SECONDARY OUTCOMES:
The anterior chamber cell score was compared between baseline and Days 3 and 7.
The total symptom score (sum of eye pain, photophobia, blurred
vision, foreign body sensation and lacrimation scores) and total
sign score (sum of anterior chamber cell, anterior chamber flare,
ciliary hyperemia, keratic precipitate and synechia of iris and
posterior scores) were compared between baseline and Days 3, 7
and 14.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeaki Ono, Principal Investigator — Department of Ophthalmology and Visual Science, Graduate School of Medicine, Hokkaido University